CLINICAL TRIAL: NCT00402298
Title: MDMA-assisted Therapy in Twelve People With War and Terrorism-related Posttraumatic Stress Disorder (PTSD)
Brief Title: Randomized Placebo-controlled Study of MDMA-assisted Therapy in People With PTSD - Israel
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated after enrolling five subjects due to staff turnover and its effects on quality of data collection.
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-3
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; MDMA; therapy; Posttraumatic stress disorder; Israel
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Full dose (125 mg) MDMA-assisted therapy (Experimental): Participants will receive an initial dose of 125 mg midomafetamine HCl followed 2.5 hours later by a supplemental dose of 62.5 mg midomafetamine HCl during the course of two day-long therapy sessions.
  Interventions: Drug: Full Dose Midomafetamine HCl
- Active Comparator (25 mg) MDMA-assisted therapy (Active Comparator): Participants will receive an initial dose of 25 mg midomafetamine HCl followed 2.5 hours later by a supplemental dose of 12.5 mg midomafetamine HCl during the course of two day-long therapy sessions.
  Interventions: Drug: Low Dose Midomafetamine HCl

INTERVENTIONS:
Drug: Full Dose Midomafetamine HCl — Participants will receive an initial dose of 125 mg midomafetamine HCl orally followed 2.5 hours later by 62.5 mg midomafetamine HCl orally during the course of a day-long therapy session.
  Other Names: midomafetamine; 3,4-methylenedioxymethamphetamine; MDMA HCl; MDMA
  Arms: Full dose (125 mg) MDMA-assisted therapy
Drug: Low Dose Midomafetamine HCl — Participants will receive an initial dose of 25 mg midomafetamine HCl orally followed 2.5 hours later by a supplemental dose of 12.5 mg midomafetamine HCl orally during the course of each of two day-long therapy sessions.
  Other Names: midomafetamine; 3,4-methylenedioxymethamphetamine; MDMA HCl; MDMA
  Arms: Active Comparator (25 mg) MDMA-assisted therapy

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy can treat PTSD in participants with PTSD. Researchers will compare two sessions of MDMA-assisted therapy with two sessions of low dose (active placebo) MDMA-assisted therapy to determine if MDMA-assisted therapy is safe and works to treat PTSD symptoms.

Participants will be randomly assigned to receive either the full dose of MDMA or low active placebo dose of MDMA during each of two experimental sessions. PTSD symptoms will be measured throughout the study.

DETAILED DESCRIPTION:
This study will examine whether two six to eight-hour long sessions of 3,4-methylenedioxymethamphetamine (MDMA)-assisted therapy scheduled two to four weeks apart are safe, and whether combining a fully therapeutic dose of MDMA with psychotherapy, compared with a low ("active placebo") dose of MDMA, will reduce PTSD symptoms, with symptoms measured four times, once at baseline and again 2, 6, and 12 months after the second experimental session. People who received the active placebo dose of MDMA can then take part in an "open label" study continuation, with the participant receiving a fully active dose of MDMA on two more six to eight hour-long psychotherapy sessions. Open-label means that the participants and the researchers know that the participant will receive the fully active dose of MDMA. People who take part in the open label study continuation have their PTSD symptoms checked six and 12 months after the second open label MDMA-assisted session.

This study will look at MDMA-assisted therapy in 12 individuals aged 18 years or older, with PTSD symptoms not improving after trying at least one treatment. At least two-thirds of participants will have diagnosed PTSD arising from war or terrorism-related trauma. Eight of 12 participants will be assigned to receive the full dose of MDMA, and four will be assigned to receive a low or "active placebo" dose of MDMA during each of two experimental sessions. The fully active dose consists of an initial dose of 125 mg MDMA HCl and a supplemental dose of 62.5 mg given 2 to 2.5 hours later. The active placebo dose consists of an initial dose of 25 mg MDMA HCl and a supplemental dose of 12.5 mg.

The study will will include two sixty minute long introductory therapy sessions, two active placebo or fully active dose MDMA-assisted therapy sessions, a sixty to ninety minute long therapy session 24 hours after each experimental session, and one to two hour-long therapy sessions occurring weekly between the first and second experimental session, and between the second experimental session and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Posttraumatic stress disorder still remaining after at least one treatment, with treatment including psychotherapy or pharmacotherapy. At least two-thirds of participants will have PTSD as a result of war and terrorism
* May meet criteria for a mood disorder.
* Must be at least 18 years old.
* Must be able to stop taking psychiatric medication from the start of the study until the two-month follow-up.
* May continue seeing an outside therapist during the study, but cannot increase the length or frequency of treatments.
* Must be able to follow all the rules and instructions relating to the experimental session, including restrictions on food and substance (alcohol and drug) consumption
* Must be willing to stay overnight in the clinic after each experimental session until the non-drug session occurring the next morning.
* Must be willing to be contacted by one of the researchers on a daily basis for a week after each experimental session.
* If a woman of childbearing potential, must have a negative pregnancy test and must agree to use an effective form of birth control.
* Must be able to speak and read Hebrew.

Exclusion Criteria:

* Cannot have history of or be diagnosed with psychotic disorder or bipolar affective disorder - 1.
* Cannot be diagnosed with dissociative identity disorder, an eating disorder with active purging, or borderline personality disorder.
* Cannot have evidence or history of significant hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder. (People with hypothyroidism who are on adequate and stable thyroid replacement will not be excluded).
* Cannot have uncontrolled hypertension, peripheral vascular disease, hepatic disease (with or without abnormal liver enzymes), or history of hyponatremia or hyperthermia.
* Cannot weigh less than 50 or more than 105 kg.
* Cannot have used "Ecstasy" more than five times during lifetime or in the past six months.
* Cannot present a serious suicide risk or be likely to require hospitalization during the course of the study.
* Cannot require ongoing concomitant therapy with a psychotropic drug.
* Cannot meet DSM-IV criteria for substance abuse or dependence for any substance save caffeine or nicotine in the past 60 days.
* Unable to give adequate consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-05-27 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2010-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Kotler, Principal Investigator — Director of Psychiatry, Beer Yaakov Mental Health Center
Locations (1):
- Be'er Ya'akov Mental Health Center, Be’er Ya‘aqov, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- Full Dose (125 mg): Participants will receive an initial dose of 125 mg MDMNA followed 2.5 hours later by a supplemental dose of 62.5 mg MDMA during the course of two day-long psychotherapy sessions.
  3,4-methylenedioxymethemphetmaine (MDMA_: Participants will receive an initial dose of 125 mg MDMA orally followed 2.5 hours later by 62.5 mg MDMA orally during the course of a day-long psychotherapy session.
- Low Dose (25 mg): 25 and 12.5 mg MDMA
  3,4-methylenedioxymethamphetamine: Participants will receive an initial dose of 25 mg MDMA orally followed 2.5 hours alter by a supplemental dose of 12.5 mg MDMA orally during the course of each of two day-long psychotherapy sessions.
Period: Overall Study
Arm/Group | Full Dose (125 mg) | Low Dose (25 mg)
Started | 3 | 2
Completed | 2 | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated after enrolling five subjects due to staff turnover and its effects on quality of data collection. Limited data was reported to the sponsor and its quality could not be assured. We have updated the record to reflect the limited data received.
Groups:
- Active Comparator (25 mg): 25 and 12.5 mg MDMA
  3,4-methylenedioxymethamphetamine: Participants will receive an initial dose of 25 mg MDMA orally followed 2.5 hours alter by a supplemental dose of 12.5 mg MDMA orally during the course of each of two day-long psychotherapy sessions.
- Total: Total of all reporting groups
Arm/Group | Full Dose (125 mg) | Active Comparator (25 mg) | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: Years] | 45.6 [32 to 66] | 39 [36 to 42] | 43 [32 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Israel | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) at 2-Month Follow-Up
Description: The Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-IV. It contains symptom subscales, a CAPS-IV total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline to two months after second MDMA-assisted experimental session
Population: One Full Dose participant did not complete a CAPS-IV assessment at the 2-month endpoint and is accordingly not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Full Dose (125 mg) MDMA-assisted Therapy: Participants will receive an initial dose of 125 mg midomafetamine HCl followed 2.5 hours later by a supplemental dose of 62.5 mg midomafetamine HCl during the course of two day-long psychotherapy sessions.
- Low Dose (25 mg) MDMA-assisted Therapy: Participants will receive an initial dose of 25 mg midomafetamine HCl orally followed 2.5 hours alter by a supplemental dose of 12.5 mg midomafetamine HCl orally during the course of each of two day-long psychotherapy sessions.
Arm/Group | Full Dose (125 mg) MDMA-assisted Therapy | Low Dose (25 mg) MDMA-assisted Therapy
Number analyzed (Participants) | 2 | 2
units on a scale | -0.5 (4.95) | -7 (18.38)

2. Secondary Outcome: Change in Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) at 6-Month Follow-Up
Description: as for outcome 1
Time Frame: Baseline to six months after second MDMA-assisted experimental session
Population: One Full Dose participant and one Low Dose participant did not complete a 6-month CAPS-IV assessment and are accordingly not included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Dose (125 mg) MDMA-assisted Therapy | Low Dose (25 mg) MDMA-assisted Therapy
Number analyzed (Participants) | 2 | 1
score on a scale | -0.5 (6.36) | 6

3. Secondary Outcome: Change in Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) at 12-month Follow-up
Description: as for outcome 1
Time Frame: Baseline to twelve months after second MDMA-assisted experimental session
Population: This study was terminated after enrolling five subjects due to staff turnover and its effects on quality of data collection. Limited data were reported to the sponsor and its quality could not be assured. All available data are reported; 12 month follow-up data available in 2 Full Dose participants, no 12 month follow-up data available in Low Dose participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Dose (125 mg) | Low Dose (25 mg)
Number analyzed (Participants) | 2 | 0
score on a scale | -7.5 (13.43) |

ADVERSE EVENTS:
Time Frame: From informed consent to study termination after 12 month follow up
Description: This study was terminated after enrolling five subjects due to staff turnover and its effects on quality of data collection. Limited data were reported to the sponsor and its quality could not be assured and therefore not analyzed.
Groups:
- Full Dose (125 mg) MDMA-assisted Therapy: Participants will receive an initial dose of 125 mg MDMNA followed 2.5 hours later by a supplemental dose of 62.5 mg MDMA during the course of two day-long psychotherapy sessions.
  3,4-methylenedioxymethemphetmaine (MDMA_: Participants will receive an initial dose of 125 mg MDMA orally followed 2.5 hours later by 62.5 mg MDMA orally during the course of a day-long psychotherapy session.
- Low Dose (25 mg) MDMA-assisted Therapy: 25 and 12.5 mg MDMA
  3,4-methylenedioxymethamphetamine: Participants will receive an initial dose of 25 mg MDMA orally followed 2.5 hours alter by a supplemental dose of 12.5 mg MDMA orally during the course of each of two day-long psychotherapy sessions.
Arm/Group | Full Dose (125 mg) MDMA-assisted Therapy | Low Dose (25 mg) MDMA-assisted Therapy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Dose (125 mg) MDMA-assisted Therapy (N=3) | Low Dose (25 mg) MDMA-assisted Therapy (N=2)
Fasciculation (Musculoskeletal and connective tissue disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Myoclonus (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated after enrolling five subjects due to staff turnover and its effects on quality of data collection. Limited data were reported to the sponsor and its quality could not be assured and therefore analysis is limited to descriptive statistics of available data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2009-04-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT00402298/ICF_000.pdf